CLINICAL TRIAL: NCT03672227
Title: Obesity Prevention in Low-Income Preschoolers: Testing the Impact of an Alternative Meal Service Approach in Head Start
Brief Title: Obesity Prevention in Head Start
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Pennington Biomedical Research Center (Other); Michigan State University (Other)
Responsible Party: Principal Investigator, Katherine Bauer, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00138002
Record Dates: First submitted 2018-09-07; First posted 2018-09-14 (Actual); Results first posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-11

CONDITIONS: Childhood Obesity
Keywords: Head Start; Family Style Dining
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: There are two arms in this study. In the intervention arm, teachers will receive the Mealtime Matters training about child nutrition. In the control arm, the teachers do not receive the Mealtime Matters until the completion of the study.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mealtime Matters Training (Experimental): This group of teachers will get a 3 hour nutrition training, followed by 2 one hour booster sessions.
  Interventions: Behavioral: Mealtime Matters Training
- Family Style Dining in Head Start (No Intervention): This group of teachers will not get the 3 hour nutrition training until the study has concluded.

INTERVENTIONS:
Behavioral: Mealtime Matters Training — This training will address common issues that Head Start teachers including how to deal with picky eaters, in addition to education about the nutritional needs of pre-school aged children.
  Arms: Mealtime Matters Training

SUMMARY:
Family style dining is a widely-advocated approach by which to feed children in early education settings. While family-style dining is hypothesized to allow children to attend to their hunger and satiety and consume only the amount of food they need to meet their energy needs, children's ability to self-regulate eating in this setting is dependent on a number of factors including early life experiences, the feeding strategies caregivers use during meals, and the eating environment. The goal of this study is to develop and implement a novel curriculum for childcare providers, Mealtime Matters, that addresses the factors that interfere with children's self-regulation of eating and offers caregivers strategies to reduce exposures that promote over-eating in the early education environment. Mealtime Matters will be pilot tested through a randomized controlled trial design with 7 Head Start classrooms, enrolling approximately 72 low-income preschool-aged children. Intervention feasibility and acceptability will be examined, as well as changes in caregiver/child mealtime interactions and children's dietary intake during meals at Head Start. Study results will inform the development of a fully-scaled efficacy trial.

DETAILED DESCRIPTION:
Obesity disproportionately affects low-income children. Already by age 5, 20% of low-income children in the US are obese, a prevalence three times higher than among high-income children. Obesity that emerges by this young age is persistent and contributes to sustained obesity and obesity-related chronic disease in adulthood. Identifying effective approaches to prevent obesity among young, low-income children is a national priority.

Family-style dining, in which children serve themselves food and drinks from communal dishes, is advocated as a strategy to prevent childhood obesity. It is theorized that family-style dining allows children to attend to their hunger and satiety, and consume only the amount of food they need to meet their energy needs. The alternative, where adults direct children's intake, is theorized to interfere with children's ability to self-regulate their eating and cause excess weight gain. Based on this theoretical model, the USDA's Child and Adult Care Food Program (CACFP), which provides meals to 4.2 million low-income children annually, and Head Start, the federally-funded preschool program that serves 42% of all preschool-aged children in poverty nationally, strongly encourage family-style dining.

Contrary to current beliefs however, the investigators posit that many low-income children are not able to self-regulate their eating and overeat when allowed to self-serve, leading to excess weight gain. Thus, family-style dining may increase, rather than decrease, obesity among low-income children. Basic behavioral and epidemiologic research suggests that chronic stress, which many low-income children experience, contributes to obesity-promoting appetite characteristics among children. Laboratory-based experiments have demonstrated that appetite characteristics such as these lead to excessive consumption when children are allowed to self-serve. Among low-income preschoolers, one-third to one-half of children consume calories in excess of Institute of Medicine recommendations during family-style meals. This excessive energy intake is driven by intake of meat and grains, while intake of nutrient-dense, lower calorie fruits and vegetables is far below recommendations. Children's excessive and unbalanced eating during family-style dining is often noted by teachers, who are uncertain how limit these behaviors.

Changing environmental supports for eating may be particularly important for modifying the dietary intake of young children who, unlike adolescents and adults, do not yet have the cognitive capacity to inhibit intake of highly palatable foods in favor of selecting food based on healthfulness. Therefore, the objective of this Collaborative Research pilot study is to conduct T2 translational research among low-income preschool children by developing an easily-implemented curriculum to support family-style dining in Head Start called Mealtime Matters, where teachers receive focused training on preschooler nutrition, appropriate portion sizes for preschool children, responsive feeding strategies, and improvements to the classroom environment that promote children's self-regulation of eating. The feasibility and potential impact of Mealtime Matters will be examined with 72 children from up to 7 Head Start classrooms in Adrian, Michigan. The investigators hypothesize that Mealtime Matters will be feasible and acceptable to teachers. Further, by reducing prompts to over-consume and empowering teachers to direct children to serve appropriate portion sizes while using responsive feeding approaches, the investigators will: 1. Increase the proportion of children consuming within an acceptable range of the recommended kilocalories (kcal) during meals at Head Start and 2. Increase the servings of fruits and vegetables children consume during meals at Head Start. Sustained engagement in these dietary behaviors can prevent excessive weight gain and obesity.

The specific aims of this trial are:

Aim 1: Examine the effect of Mealtime Matters on children's dietary intake during meals at Head Start.

Aim 2: Examine the effect of Mealtime Matters on teacher/child mealtime interactions at Head Start.

Aim 3: Determine the feasibility and acceptability of Mealtime Matters among Head Start teachers.

ELIGIBILITY:
TEACHERS

Inclusion Criteria:

- employed as teachers in the Adrian Public School's Head Start Program

Exclusion Criteria:

- N/A

CHILDREN

Inclusion Criteria:

* enrolled in the Adrian Public School's Head Start Program
* the specific age range for children selected of 3-4 years by September 1 of the given academic year is based on the age of eligibility for Head Start enrollment
* the custodial and legal guardian is able to provide valid consent

Exclusion Criteria:

* child has serious medical problems
* the child is a foster child

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-08-24 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine W Bauer, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants include teachers, children within the classrooms of these teachers, and a parent of each child. Milestones used to break out number in each group enrolled.
Groups:
- Family Style Dining in Head Start: This group of teachers will not get the nutrition training until the study has concluded.
Period: Overall Study
Arm/Group | Mealtime Matters Training | Family Style Dining in Head Start
Started | 112 | 52
Teachers Started | 8 | 6
Children Started | 52 | 23
Parents Started | 52 | 23
Completed | 105 | 52
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mealtime Matters Training | Family Style Dining in Head Start | Total
Number analyzed (Participants) | 112 | 52 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 53 | 23 | 76
  Between 18 and 65 years | 59 | 28 | 87
  >=65 years | 0 | 1 | 1
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22.4 [3.6 to 30.8] | 23.6 [3.7 to 29.2] | 23.3 [3.6 to 30.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 41 | 120
  Male | 33 | 11 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 19 | 48
  Not Hispanic or Latino | 83 | 33 | 116
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 8 | 25
  White | 78 | 41 | 119
  More than one race | 11 | 1 | 12
  Unknown or Not Reported | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 112 | 52 | 164

OUTCOME MEASURES:

1. Primary Outcome: Change in Percentage of Children Over-consuming Energy During Lunch Attributable to Mealtime Matters
Description: Dietary intake data will be collected via the Remote Food Photography Method over 2 lunches at Head Start among children in intervention and control classrooms to identify the proportion of children over-consuming energy during meals. Over-consumption is defined as an average per meal intake > 332 kilocalories based on IOM recommendations regarding median energy intake recommended for 3 to 5 year olds' lunch in CACFP settings.
Time Frame: baseline, 6 weeks post-intervention
Population: Only children were included in this analysis.
Measure: Number; unit: Percent of Participants
Arm/Group | Mealtime Matters Training | Family Style Dining in Head Start
Number analyzed (Participants) | 46 | 23
Percent of Participants | -10.9 | -56.5

2. Secondary Outcome: Change in Teachers' Feeding Practices Attributable to Mealtime Matters
Description: Data will be collected at baseline among teachers in intervention and control classrooms. Two lunch periods will be video and audio recorded to identify teachers' feeding practices.
Time Frame: baseline, 6 weeks post-intervention
Population: No data was collected from video and audio recordings due poor inter-rater reliability of trained coders.
Arm/Group | Mealtime Matters Training | Family Style Dining in Head Start
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Teachers Satisfied With Mealtime Matters [ Time Frame: Post-training ]
Description: Data on teacher satisfaction will be collected via teacher questionnaires immediately post training to better understand whether the teachers found the training interesting, relevant, easy to implement, and useful.
Time Frame: 3 hours
Population: Teachers who completed the 3-hour nutrition training
Measure: Count of Participants; unit: Participants
Arm/Group | Mealtime Matters Training | Family Style Dining in Head Start
Number analyzed (Participants) | 7 | 0
Participants | 7 | 0

4. Secondary Outcome: Number of Teachers Satisfied With Mealtime Matters
Description: Data on teacher satisfaction will be collected via teacher questionnaires post-intervention to better understand whether the teachers found the training interesting, relevant, easy to implement, and useful.
Time Frame: 6 weeks post-intervention
Population: Teachers assigned to Mealtime Matters Training
Measure: Count of Participants; unit: Participants
Arm/Group | Mealtime Matters Training | Family Style Dining in Head Start
Number analyzed (Participants) | 8 | 0
Participants | 8 |

ADVERSE EVENTS:
Time Frame: From baseline to 6-weeks post intervention follow up
Arm/Group | Mealtime Matters Training | Family Style Dining in Head Start
All-Cause Mortality (participants affected / at risk) | 0/112 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/52
Other Adverse Events (participants affected / at risk) | 0/112 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT03672227/Prot_SAP_000.pdf